CLINICAL TRIAL: NCT01990690
Title: Role of Antioxidants in Unexplained Oligohydramnios,A Randomized Trial
Acronym: ao&uoh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, Assistant professor ob/gyn, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aouoh
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Oilgohydramnios
Keywords: oligohydramnios,antioxidant,oxidative stress and pregnancy outcomes
MeSH Terms: conditions — Oligohydramnios | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti oxidant omega 3 (Active Comparator): The patients were randomized to receive either a daily dose of omega-3 plus as antioxidant once daily for two weeks or a daily placebo then stored in envelopes numbered from 1 to 140
  Interventions: Drug: anti oxidant omega 3
- placebo (Placebo Comparator): Group 1 was given omega -3 plus (Sedico medical company) as antioxidant once daily for two weeks.
  Group 2 was given a placebo once daily for two weeks.
  Interventions: Drug: anti oxidant omega 3

INTERVENTIONS:
Drug: anti oxidant omega 3 — Soft gelatineous capsule (Sedico medical company) each capsule contains:
  * Fish oil (30) % (Eicosapentaenoic acid (EPA) 18 % / Docosahexaenoic acid (DHA) 12 % ) natural source of Omega 3 Fatty acids.
  * Wheat germ oil (Tocopherol: N.N.T. 0.22 %) which is rich and natural source of Vitamin E (protects the oils from oxidation. besides its well known that requirements of vitamin E increases with increased dietary amounts of polyunsaturated fatty acids).
  Group 1 was given omega -3 plus (Sedico medical company) as antioxidant once daily for two weeks.
  Other Names: omega 3 plus

SUMMARY:
To predict the effect of antioxidants in cases of oligohydramnios

DETAILED DESCRIPTION:
Type of study:

This is a prospective randomized controlled study that was done in department of obstetrics and gynecology of Assiut University Hospital.

Aim of the work:

1. To study the effect of antioxidants in cases of oligohydramnios.
2. To study the effect of antioxidants on mode of delivery and neonatal outcome.
3. To commence special recommendations from the study about the use of antioxidants in cases of oligohydramnios of unknown cause and cases of oligohydramnios associated with pregnancy induced hypertension.

Inclusion criteria:

Patients with gestational age between 30-34 weeks with:

* Oligohydramnios of unknown cause.
* Oligohydramnios assosiatd with Pregnancy induced hypertension (PIH).

Exclusion criteria:

1. Premature rupture of membranes.
2. Oligohydramnios in postdates pregnancy (>41 weeks).
3. Fetal anomalies.
4. IUGR.
5. Patients using non steroidal anti-inflammatory drugs.

Assessment of the patients:

The target population was assessed to find the participating women suitable for the study, this assessment was done to verify inclusion criteria and to exclude any women has any of the exclusion criteria.

Ultrasongraphic evaluation:

Ultrasongraphy was done for estimation of amniotic fluid index by measuring the vertical diameter of the pockets of amniotic fluid in four sections of the uterus and add them together. This gives them a number known as amniotic fluid index (AFI). If the AFI is less than 5 centimeters, the pregnant woman has oligohydramnios

Composition of omega-3 plus:

Soft gelatineous capsule (Sedico medical company) each capsule contains:

* Fish oil (30) % (Eicosapentaenoic acid (EPA) 18 % / Docosahexaenoic acid (DHA) 12 % ) natural source of Omega 3 Fatty acids.
* Wheat germ oil (Tocopherol: N.N.T. 0.22 %) which is rich and natural source of Vitamin E (protects the oils from oxidation. besides its well known that requirements of vitamin E increases with increased dietary amounts of polyunsaturated fatty acids).

ELIGIBILITY:
Inclusion Criteria:

* Patients with gestational age between 30-34 weeks with:
* Oligohydramnios of unknown cause.

Exclusion Criteria:

* 1- Premature rupture of membranes. 2- Oligohydramnios in postdates pregnancy (>41 weeks). 3- Fetal anomalies. 4- IUGR. 5- Patients using non steroidal anti-inflammatory drugs. 6 - Oligohydramnios assosiatd with Pregnancy induced hypertension (PIH).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
improvement of amniotic fluid index | 4 weeks
  Treatment was started immediately and continued for two weeks. The patients were randomized to receive either a daily dose of omega-3 plus as antioxidant once daily for two weeks or a daily placebo then stored in envelopes numbered from 1 to 140. The envelopes were numbered and randomized according to computer-generated randomization tables to ensure an equal number of patients in each arm. Throughout the trial, access to the randomization code was available only to the pharmacist who manufactured the placebo and packed the envelopes and was not available to any of the treating physicians or patients.

SECONDARY OUTCOMES:
The changes in Doppler resistance index | 4 weeks
  The resistance index is measured in the uterine and umbilical artery by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M D, Principal Investigator — Women's Health Hospital
Locations (1):
- Women's Health Hospital, Asyut, Egypt